CLINICAL TRIAL: NCT02647489
Title: Safety and Immunogenicity of the Placental Malaria Vaccine Candidate PAMVAC Adjuvanted With Alhydrogel, GLA-SE or GLA-LSQ in Healthy Malaria-Naïve Adults and Healthy, Lifelong Malaria-Exposed, Nulligravid Adult Women
Brief Title: Safety and Immunogenicity of the Placental Malaria Vaccine Candidate PAMVAC Variously Adjuvanted
Acronym: PAMVAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University of Copenhagen (Other); Université d'Abomey-Calavi (Other); European Vaccine Initiative (Other); Institut de Recherche pour le Developpement (Other Government); ExpreS2ion Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PAMVAC1_15
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2016-10

CONDITIONS: Malaria, Antepartum
MeSH Terms: conditions — Malaria | interventions — Aluminum Hydroxide; glucopyranosyl lipid-A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- 1A - 20 µg PAMVAC + Alhydrogel (Experimental): The study participant will get 20 µg of PAMVAC adjuvanted with Alhydrogel administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: Alhydrogel
- 2A - 20 µg PAMVAC + GLA-SE (Experimental): The study participant will get 20 µg of PAMVAC adjuvanted with GLA-SE administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: GLA-SE
- 3A - 20 µg PAMVAC + GLA-LSQ (Experimental): The study participant will get 20 µg of PAMVAC adjuvanted with GLA-LSQ administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: GLA-LSQ
- 4A - 50 µg PAMVAC + Alhydrogel (Experimental): The study participant will get 50 µg of PAMVAC adjuvanted with Alhydrogel administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: Alhydrogel
- 5A - 50 µg PAMVAC + GLA-SE (Experimental): The study participant will get 50 µg of PAMVAC adjuvanted with GLA-SE administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: GLA-SE
- 6A - 50 µg PAMVAC + GLA-LSQ (Experimental): The study participant will get 50 µg of PAMVAC adjuvanted with GLA-LSQ administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: GLA-LSQ
- 1B - 50 µg PAMVAC + Alhydrogel (Experimental): The study participant will get 50 µg of PAMVAC adjuvanted with Alhydrogel administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: Alhydrogel
- 2B - 50 µg PAMVAC + GLA-SE (Experimental): The study participant will get 50 µg of PAMVAC adjuvanted with GLA-SE administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: GLA-SE
- 3B - 100 µg PAMVAC + Alhydrogel (Experimental): The study participant will get 100 µg of PAMVAC adjuvanted with Alhydrogel administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: Alhydrogel
- 4B - 100 µg PAMVAC + GLA-SE (Experimental): The study participant will get 100 µg of PAMVAC adjuvanted with GLA-SE administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Biological: PAMVAC; Biological: GLA-SE
- 5B - Placebo (Placebo Comparator): The study participant will get Placebo (physiological saline solution) administrated three times with each time 28 days interval (day 0-28-56)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PAMVAC
  Arms: 1A - 20 µg PAMVAC + Alhydrogel; 1B - 50 µg PAMVAC + Alhydrogel; 2A - 20 µg PAMVAC + GLA-SE; 2B - 50 µg PAMVAC + GLA-SE; 3A - 20 µg PAMVAC + GLA-LSQ; 3B - 100 µg PAMVAC + Alhydrogel; 4A - 50 µg PAMVAC + Alhydrogel; 4B - 100 µg PAMVAC + GLA-SE; 5A - 50 µg PAMVAC + GLA-SE; 6A - 50 µg PAMVAC + GLA-LSQ
Biological: Alhydrogel
  Arms: 1A - 20 µg PAMVAC + Alhydrogel; 1B - 50 µg PAMVAC + Alhydrogel; 3B - 100 µg PAMVAC + Alhydrogel; 4A - 50 µg PAMVAC + Alhydrogel
Biological: GLA-SE
  Arms: 2A - 20 µg PAMVAC + GLA-SE; 2B - 50 µg PAMVAC + GLA-SE; 4B - 100 µg PAMVAC + GLA-SE; 5A - 50 µg PAMVAC + GLA-SE
Biological: GLA-LSQ
  Arms: 3A - 20 µg PAMVAC + GLA-LSQ; 6A - 50 µg PAMVAC + GLA-LSQ
Other: Placebo
  Arms: 5B - Placebo

SUMMARY:
Despite having developed robust acquired immunity against complications of malaria, women can return to a susceptible state during their first pregnancies and contribute significantly to the burden of severe malaria in highly endemic areas. Naturally acquired protection against placental malaria correlates with the presence of high concentration of immunoglobulin G molecules (IgGs) against VAR2CSA, a parasite protein of the var gene family that is essential for the binding of infected erythrocytes to CSA in the placenta.

To induce high concentrations of specific IgGs, subjects will receive escalating doses of PAMVAC vaccine antigen adjuvanted with Alhydrogel, Glucopyranosyl Lipid Adjuvant-Stable Emulsion (GLA-SE) or Glucopyranosyl Lipid Adjuvant-Liposome-QS-21 Formulation (GLA-LSQ). Three injections with the same dosage and adjuvant will be done, each 28 days apart (Day 0, 28 and 56). Control subjects will receive physiological saline instead of the vaccine and dose escalation will be staggered to ensure safety during the trial.

DETAILED DESCRIPTION:
Phase 1, staggered, two-center, dose-escalation trial. The trial will be conducted in two stages. The first in Germany (first in man and dose escalation) and the second in a malaria-endemic area in the target group (randomized, controlled, dose-finding).

First in man administration and dose escalation from 20 to 50 μg per injection of PAMVAC adjuvanted with Alhydrogel, GLA-SE and GLA-LSQ will be done in healthy, malaria-naïve adults in Germany (Stage 1).

Subsequently, PAMVAC will be administered to healthy, lifelong malaria-exposed nulligravid women in Benin at doses of 50 and 100 μg, adjuvanted with Alhydrogel and GLA-SE (Stage 2).

The PAMVAC vaccine is a VAR2CSA protein-based vaccine, aiming to protect fetus and mother against the adverse effects of placental malaria during pregnancy. As the interaction between the parasite protein VAR2CSA and CSA in the human placenta is a key element in the pathogenesis of placental malaria, a vaccine should elicit the type of immunoglobulins that block the binding of VAR2CSA to CSA. A small sub-unit of the VAR2CSA protein (ID1-ID2a) has been selected as the PAMVAC vaccine antigen. In animal models IgGs induced by immunization with the recombinant PAMVAC antigen are able to inhibit homologous parasite-infected erythrocyte adhesion to CSA in vitro.

The three adjuvants are Alhydrogel, an aluminum hydroxide gel widely used as adjuvant in this trial; GLA-SE and GLA-LSQ, synthetic TLR-4 agonists with a strong immune stimulatory effect formulated either in a stable oil-in-water emulsion (SE) or together with QS-21 (Saponin derived from the Quillaja saponaria tree) as liposome (LSQ).

In Benin, one group will receive a placebo control (physiological saline). Allocation to placebo, PAMVAC+Alhydrogel or PAMVAC+GLA-SE, will be randomized and the trial team as well as the participants will be kept blinded (double-blinded) to their allocation.

All participants (Stage 1+2) will receive three intramuscular injections in four-week intervals.

Each dose-escalation is conditional on a positive safety assessment by an independent Safety Monitoring Board (SMB) and sponsor approval. One individual of each PAMVAC-adjuvant combination will serve as sentinel. The sentinel will be injected one day before the rest of the group.

There will be a minimum of 4 weeks stagger between the first immunization of Groups 1A-3A and Groups 4A-6A.

Group 1A (n = 3) - 20 µg PAMVAC+Alhydrogel Group 2A (n = 3) - 20 µg PAMVAC+GLA-SE Group 3A (n = 3) - 20 µg PAMVAC+GLA-LSQ Group 4A (n = 9) - 50 µg PAMVAC+Alhydrogel Group 5A (n = 9) - 50 µg PAMVAC+GLA-SE Group 6A (n = 9) - 50 µg PAMVAC+GLA-LSQ

Following safety assessment by the SMB after the first dose in Groups 4A-6A and approval by the sponsor, Stage 2 (in Benin) will be initiated. Here, the target population of PAMVAC (healthy nulligravid women in a malaria-endemic area) will be vaccinated. Upon SMB review and approval by the sponsor Groups 1B-2B and half the subjects from the control Group 5B will receive vaccinations. One participant allocated to group 1B, 2B and 5B will receive the first immunization at least one day before the rest of the group.

Group 1B (n=9) - 50 µg PAMVAC+Alhydrogel Group 2B (n=9) - 50 µg PAMVAC+GLA-SE Group 3B (n=3) - 100 µg PAMVAC+Alhydrogel Group 4B (n=3) - 100 µg PAMVAC+GLA-SE Group 5B (n=6) - Placebo (physiological saline solution)

There will be a 4 weeks stagger between Groups 1B-2B and Group 3B-4B and the remaining subjects of the control Group 5B to allow for safety evaluation by the SMB. Here, the same system of sentinel vaccination as for the lower dose will be used; one participant allocated to group 3B, 4B and 5B will receive the first immunization at least one day before the rest of the group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged 18-45 years.
* Able and willing (in the investigator's opinion) to comply with all trial requirements.
* General good health based on history and clinical examination
* Written informed consent
* Women only: Must agree to practice continuous effective contraception for the duration of the trial (a method which results in a low failure rate; i.e. less than 1% per year). Women will be counseled about effective contraception methods and, if required, can be provided with adequate contraceptives by the investigator team.
* Available to participate in follow up for the duration of trial (36 weeks following first injection)
* Reachable by phone during the whole trial period

Exclusion Criteria:

* Pregnancy, lactation or intention to become pregnant during the trial
* Previous participation in a malaria vaccine trial
* HIV infection
* Any confirmed or suspected immunosuppressive or immunodeficient state, asplenia, recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* Presence of autoimmune diseases requiring systemic treatment (e.g. rheumatic diseases)
* Use of immunoglobulins or blood products within 3 months prior to enrolment
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the trial period
* History of malaria or travel in malaria-endemic areas within the past 6 months
* Intention to travel to malaria endemic countries during the trial period
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition that may affect participation in the trial
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 60 g (men) or 40 g (women) per day or a carbohydrate deficient transferrin (CDT) level ≥2.5%
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Positive for hepatitis B surface antigen (HBs-antigen)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Known hypersensitivity to any of the vaccine components (adjuvant or peptide)
* Any clinically significant abnormal finding on biochemistry or hematology blood tests, urine analysis or clinical examination
* History of seizure, except for sporadic febrile convulsions in childhood
* Any other significant disease, disorder or finding which, in the opinion of the investigator, may significantly increase the risk to the volunteer because of participation in the trial; affect the ability of the volunteer to participate in the trial or impair interpretation of the trial data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Number and grade of adverse events (Grade 1-3 and serious adverse events) possibly, likely and definitely related to vaccination | From the first administration of the interventions through study completion, an average of 1 and a half years

SECONDARY OUTCOMES:
Area under the curve of anti-PAMVAC IgG concentration | Before first administration, 1, 4, 5, 8, 9, 12, 24 and 36 weeks after first administration

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin G Mordmüller, MD, Principal Investigator — University Hospital Tübingen; Saadou Issifou, MD, Principal Investigator — Université d'Abomey-Calavi
Locations (1):
- Institut de Recherche Clinique du Benin (IRCB), Abomey-Calavi, Benin

REFERENCES:
- [Derived] Larsen MD, Lopez-Perez M, Dickson EK, Ampomah P, Tuikue Ndam N, Nouta J, Koeleman CAM, Ederveen ALH, Mordmuller B, Salanti A, Nielsen MA, Massougbodji A, van der Schoot CE, Ofori MF, Wuhrer M, Hviid L, Vidarsson G. Afucosylated Plasmodium falciparum-specific IgG is induced by infection but not by subunit vaccination. Nat Commun. 2021 Oct 5;12(1):5838. doi: 10.1038/s41467-021-26118-w. PMID 34611164
- [Derived] Gamain B, Chene A, Viebig NK, Tuikue Ndam N, Nielsen MA. Progress and Insights Toward an Effective Placental Malaria Vaccine. Front Immunol. 2021 Feb 25;12:634508. doi: 10.3389/fimmu.2021.634508. eCollection 2021. PMID 33717176
- [Derived] Mordmuller B, Sulyok M, Egger-Adam D, Resende M, de Jongh WA, Jensen MH, Smedegaard HH, Ditlev SB, Soegaard M, Poulsen L, Dyring C, Calle CL, Knoblich A, Ibanez J, Esen M, Deloron P, Ndam N, Issifou S, Houard S, Howard RF, Reed SG, Leroy O, Luty AJF, Theander TG, Kremsner PG, Salanti A, Nielsen MA. First-in-human, Randomized, Double-blind Clinical Trial of Differentially Adjuvanted PAMVAC, A Vaccine Candidate to Prevent Pregnancy-associated Malaria. Clin Infect Dis. 2019 Oct 15;69(9):1509-1516. doi: 10.1093/cid/ciy1140. PMID 30629148